CLINICAL TRIAL: NCT02740894
Title: Can Epidermal Growth Factor Receptor - Tyrosine Kinase Inhibitor Improve the Postoperative Survivorship for Inoperable Non-small Cell Lung Cancer With Spinal Metastasis of the Thoracic and Lumbar Spine?- A Retrospective Comparison With Platinum-based Chemotherapy
Brief Title: Can Epidermal Growth Factor Receptor Improve the Postoperative Survivorship for Inoperable Non-small Cell Lung Cancer With Spinal Metastasis ?
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, ST Wang, Chief of spinal surgery. Taipei Veterans General Hospital, Taiwan, Taipei Veterans General Hospital, Taiwan
Other Study IDs: 2016-02-006CC
Record Dates: First submitted 2016-04-05; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Is Targeted Therapy Increasing Survival Inoperable Nonsmall Cell Lung Cancer With Spinal Metastasis ?
MeSH Terms: interventions — Gefitinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- targeted therapy: according to national healthy policy, targeted therapy is the optional therapy
  Interventions: Drug: Gefitinib
- traditional chemotherapy: according to national healthy policy, chemotherapy is the first line treatment.
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib
  Other Names: Targeted therapy

SUMMARY:
Not significantly increased survival in T/T

ELIGIBILITY:
Inclusion Criteria:

* NSCLC with spinal metastasis

Exclusion Criteria:

* brain metastasis and expected survival < 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: NSCLC with spinal metastasis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Survival and neurologic outcome of 60 participants receiving targeted therapy for nonsmall cell lung cancer with spinal metastaasis. Neurological outcome by Frankel grading and ambulation status. | postoperation to mortality, up to 2 year